CLINICAL TRIAL: NCT03596060
Title: Regional vs General Anesthesia in Patients With Hip Fracture Under Treatment With Clopidogrel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Aikaterini Tsiaka, MD, Consultant Anaesthesiologist, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5505/19.10.2017
Record Dates: First submitted 2018-06-02; First posted 2018-07-23 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Hip Fractures
Keywords: hip fracture, general anesthesia, regional anesthesia, clopidogrel, cognitive impairment, mortality
MeSH Terms: conditions — Hip Fractures; Cognitive Dysfunction | interventions — Fentanyl; Propofol; Rocuronium; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (Active Comparator): Hip fracture patients older or equal to 65 years of age, who receive clopidogrel, will be randomly assigned to undertake surgery under general anesthesia in the first 48 hours. Anesthetics to be used are propofol, fentanyl and rocuronium. Maintenance will be achieved with remifentanyl and propofol (TIVA) and the depth of anesthesia will be monitored by BIS. Morphine will be administered bolus IV immediately postoperatively.
  Interventions: Drug: Fentanyl; Drug: Propofol; Drug: Rocuronium; Drug: Morphine
- Regional anesthesia (Active Comparator): Hip fracture patients older or equal to 65 years of age, who receive clopidogrel, will will be randomly assigned undertake surgery under regional anesthesia (spinal) at least 5 days after the discontinuation of clopidogrel. Anesthetics to be used are chirochaine 0.5% and fentanyl.
  Interventions: Drug: Fentanyl; Drug: Chirochaine

INTERVENTIONS:
Drug: Fentanyl — Fentanyl will be used for introduction in both regional and general anesthesia. It will also be used for general anesthesia maintenance.
Drug: Propofol — Propofol will be used for introduction in general anesthesia.
  Arms: General anesthesia
Drug: Rocuronium — Rocuronium will be used for introduction in general anesthesia.
  Arms: General anesthesia
Drug: Chirochaine — Chirochaine 0.5% will be used in regional anesthesia.
  Arms: Regional anesthesia
Drug: Morphine — Morphine will be administered bolus iv in General anesthesia group postoperatively before patients leave OR.
  Arms: General anesthesia

SUMMARY:
This study compares general to regional anesthesia concerning morbidity and mortality in patients older than or equal to 65 years old who receive clopidogrel and are to be submitted in hip fracture surgery. Half of participants will receive general anesthesia the first 48 hours and the other half will receive regional anesthesia after 5 days of the discontinuation of clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than or equal to 65 years old with hip fracture
* Native language greek and capable of speaking and writing
* Primary school graduated
* Is about to undergo in orthopedic surgery
* Participants should be available until the end of the prefixed end date of the research

Exclusion Criteria:

* Severe hearing impairment and visual acuity
* Major cognitive impairment (Mini Mental State Examination <24)
* Medical history of central nervous system disease including stroke with neurological deficit
* Medical history of alcohol or drug abuse
* Dementia, Parkinson disease, Alzheimer disease
* Contraindication for general or regional anesthesia
* Severe contraindication for antiplatelet agent discontinuation
* Multiple failures
* Receiving other coagulants
* No written consent

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  To compare postoperative 30-day mortality between General anesthesia and Regional anesthesia group

SECONDARY OUTCOMES:
Major Cardiovascular Events | Events will be recorded for both groups from date of surgery postop up to 12 months or date of death from any cause, with intermediate recordings in 1, 3 and 6 months periods in survivors
  To check and compare between General anesthesia and Regional anesthesia group for major cardiovascular events (arrhythmias, stroke, cardiac arrest, acute myocardial infract, acute respiratory oedema, pulmonary embolism) postoperatively in 30 days and 3, 6, 12 months.
Change in cognitive status | Cognitive function will be measured for both groups on admission (preop), 6 months and 12 months postop
  To measure and compare, between General anesthesia and Regional anesthesia group, Cognitive status using Mini Mental State Examination and Clock Test before surgery and 6, 12 months postoperatively
Delirium | Occurrence of delirium will be measured, for both groups, on admission (preop) and days 2, 3, 4 and 7 postop (two tests per day, morning and evening hours)
  Occurrence of delirium and comparison between General anesthesia and Regional anesthesia group with the use of Confusion Assessment Method before surgery and in 2, 3, 4 and 7 days postoperatively.
Adverse events postoperatively | 30 days
  Occurrence of adverse events in both General anesthesia and Regional anesthesia groups, especially respiratory, renal, surgical trauma in 30 days postoperatively.
Re-admissions | 30 days
  Re admissions in both General anesthesia and Regional anesthesia groups in 30 days postoperatively.
Postoperative analgesic use | 30 days
  Use of analgesics (pethidine, paracetamol), counted in milligrams as a mean per day, from the time patients are transfered to the orthopedic ward until 30 days postop in both General anesthesia and Regional anesthesia groups targeting Numerical Rating Scale score <4 (range is from 0 to 10 and a higher score indicates greater pain intensity).
Time of hospitalization | Time to discharge will be considered the time duration from date of surgery until the date of discharge or date of death from any cause while hospitalised, whichever came first, assessed up to 1 month
  To check and compare in both General anesthesia and Regional anesthesia groups time to hospital discharge.
Adverse events intraoperatively | During operation time frame
  To check and compare in both General anesthesia and Regional anesthesia groups incidence of low blood pressure (< 20% from baseline), bradycardia (<50 bpm), hemorrhage and need of blood transfusions, use of antifibrinolytics intraoperatively
Functionality in daily living | 6 months
  To check and compare between both General anesthesia and Regional anesthesia groups 6 months postoperatively functionality using Instrumental Activities of Daily Living scale
Timed Up and Go Test (TUG) | Measurements will be assessed 1, 3 and 6 months postop
  To determine fall risk and measure the progress of balance, sit to stand, and walking using Timed Up and Go Test (TUG) and compare these attributes between General anesthesia and Regional anesthesia groups 1, 3 and 6 months postoperatively
EQ-5D-5L (EuroQol group, 5 dimensions, 5 levels) | Measurements will be assessed at 1, 3 and 6 months postop
  With the use of EQ-5D-5L to check and compare between General anesthesia and Regional anesthesia groups 1, 3 and 6 months postoperatively mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Oxford hip score | Measurements will be assessed at 1, 3 and 6 months postop
  To assess function and pain in both General anesthesia and Regional anesthesia groups 1, 3 and 6 months postoperatively by using Oxford hip score

CONTACTS AND LOCATIONS:
Locations (1):
- Larissa University Hospital, Larissa, Greece

IPD SHARING:
Plan to Share IPD: Undecided